CLINICAL TRIAL: NCT03283670
Title: Inhaled Nitrous Oxide for Treatment-Resistant Depression: Optimizing Dosing Strategies
Acronym: NARSAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Ben Palanca, Associate Professor of Anesthesiology and Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201608024
Record Dates: First submitted 2016-11-09; First posted 2017-09-14 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant
Keywords: Depression; treatment-resistant
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: Each participant receives the 3 inhalation types in randomized, one hour sessions separated by at least 4 weeks
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. 25% nitrous oxide, 25% nitrogen, 25% oxygen (Experimental): Participants will be studied for 14 visits over approximately 18 weeks. The participants will receive 1 hour-long gas inhalation mixtures at 3 different times, which are randomly assigned.
  Interventions: Drug: Nitrous Oxide 25%
- 2. 50% nitrous oxide, 50% oxygen (Experimental): Participants will be studied for 14 visits over approximately 18 weeks. The participants will receive 1 hour-long gas inhalation mixtures at 3 different times, which are randomly assigned.
  Interventions: Drug: Nitrous Oxide 50%
- 3. Placebo gas: 50% nitrogen(inert), 50% oxygen (Placebo Comparator): Participants will be studied for 14 visits over approximately 18 weeks. The participants will receive 1 hour-long gas inhalation mixtures at 3 different times, which are randomly assigned.
  Interventions: Drug: Placebo Gas

INTERVENTIONS:
Drug: Nitrous Oxide 25% — Nitrous oxide, an odorless, colorless gas typically used as an induction agent for general anesthesia or for dental sedation, is a known N-methyl-D-aspartate (NMDA) antagonist. It will be given at a concentration of 25% nitrous oxide/50% oxygen/25% nitrogen.
  Other Names: One hour inhalation of 25% nitrous oxide
  Arms: 1. 25% nitrous oxide, 25% nitrogen, 25% oxygen
Drug: Nitrous Oxide 50% — Nitrous oxide, an odorless, colorless gas typically used as an induction agent for general anesthesia or for dental sedation, is a known N-methyl-D-aspartate (NMDA) antagonist. It will be given at a concentration of 50% nitrous oxide/50% oxygen.
  Other Names: One hour inhalation of 50% nitrous oxide
  Arms: 2. 50% nitrous oxide, 50% oxygen
Drug: Placebo Gas — Placebo gas given at 50% nitrogen [inert]/50% oxygen.
  Other Names: One hour inhalation of placebo gas
  Arms: 3. Placebo gas: 50% nitrogen(inert), 50% oxygen

SUMMARY:
The purpose of the study aims to determine whether different concentrations of nitrous oxide (N2O) have different antidepressant effects for adults with treatment-resistant major depression.

DETAILED DESCRIPTION:
Most clinical major depression responds to standard treatments (medication and psychotherapy); however, a significant subset of depressed patients (15-20%) do not respond to these treatments and are referred to as treatment-resistant major depression (TRMD). New treatments for TRMD are needed, and one promising line of research are drugs known as N-methyl-D-aspartate (NMDA) glutamate receptor antagonists. In a recent pilot study, our group demonstrated that the NMDA antagonist nitrous oxide is effective in TRMD.

All patients will receive 3 randomized, one hour nitrous oxide inhalations to placebo (0% N2O), low dose (25% N2O), and high dose (50% N2O). Inhalation sessions will be at least 4 weeks apart. Mood will be assessed at baseline, 2 and 24 hours, and 1, 2, and 4 weeks post-inhalation for each dose.

ELIGIBILITY:
Inclusion Criteria

1. Adults 18-75 years of age;
2. Current diagnosis of unipolar major depressive disorder (MDD) without psychosis as confirmed by structured clinical interview for DSM-IV disorders;
3. A score of >= 9 on the Montgomery-Åsberg Depression Rating Scale (MADRS);
4. Documented (i.e., chart review) lifetime failure to respond to >=3 adequate dose/duration antidepressant treatment trials, ≥1 medication failure in the current depressive episode;
5. Good command of the English language.

Exclusion Criteria

1. Meets criteria for any DSM-IV diagnosis for schizophrenia, bipolar, schizoaffective, obsessive-compulsive, personality, or panic disorders;
2. Any recent (within past 12 months) history of substance dependence or abuse (except tobacco), determined by reported history or urine drug screen;
3. Ability to become pregnant and not using effective contraception;
4. Contraindication against the use of nitrous oxide:

   1. Pneumothorax
   2. Bowel obstruction
   3. Middle ear occlusion
   4. Elevated intracranial pressure
   5. Chronic cobalamin and/or folate deficiency treated with folic acid or vitamin B12
   6. Pregnant patients
   7. Breastfeeding women
5. Inability to provide informed consent;
6. Any other factor that in the investigators' judgment may affect patient safety or compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Palanca, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Derived] de Leon VC, Kumar A, Nagele P, Palanca BJ, Gott B, Janski A, Zorumski CF, Conway CR. Nitrous Oxide Reduced Suicidal Ideation in Treatment-Resistant Major Depression in Exploratory Analysis. J Clin Psychiatry. 2023 Aug 16;84(5):22br14725. doi: 10.4088/JCP.22br14725. No abstract available. PMID 37585253

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Participants: Participants will be studied for 14 visits over approximately 18 weeks. The participants will receive 1 hour-long gas inhalation mixtures at 3 different times, which are randomly assigned.
  1. 25% nitrous oxide, 25% nitrogen, 25% oxygen
  2. 50% nitrous oxide, 50% oxygen
  3. Placebo gas: 50% nitrogen(inert), 50% oxygen
Period: Placebo Gas
Arm/Group | Study Participants
Started | 24
Completed | 22
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: 25% Nitrous Oxide
Arm/Group | Study Participants
Started | 24
Completed | 20
Not Completed | 4
Not completed — Withdrawal by Subject | 4
Period: 50% Nitrous Oxide
Arm/Group | Study Participants
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 44 [26 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression Symptoms Measured by the Hamilton Depression Rating Scale- 21 Items
Description: Change in depression symptoms measured by the Hamilton Depression Rating Scale- 21 items. The HAMD-21 is designed to rate the severity of depression in patients. Although it contains 21 areas, calculate the patient's score as the total score on the first 17 answers. Scale: 0=absent, 4=worst level possible) the scores on the individual items are summed. Changes will be based on measurements obtained at baseline, approximately 2 hours after inhalation, and approximately 24 hours after inhalation. Changes are based on subtracti on of baseline score.
Time Frame: 2 and 24 hours after inhalation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 25% Nitrous Oxide: 25% nitrous oxide, 25% nitrogen, 25% oxygen. Participants will be studied for 14 visits over approximately 18 weeks. The participants will receive 1 hour-long gas inhalation mixtures at 3 different times, which are randomly assigned.
- 50% Nitrous Oxide: 50% nitrous oxide, 50% oxygen. Participants will be studied for 14 visits over approximately 18 weeks. The participants will receive 1 hour-long gas inhalation mixtures at 3 different times, which are randomly assigned.
- Placebo Gas: 50% nitrogen(inert), 50% oxygen. Participants will be studied for 14 visits over approximately 18 weeks. The participants will receive 1 hour-long gas inhalation mixtures at 3 different times, which are randomly assigned.
Arm/Group | 25% Nitrous Oxide | 50% Nitrous Oxide | Placebo Gas
Number analyzed (Participants) | 20 | 23 | 22
score on a scale
  2 Hours | -3.0 (3.9) | -3.8 (4.30) | -3.9 (4.3)
  24 Hours | -4.0 (6.6) | -5.5 (5.8) | -6.0 (6.4)
Statistical Analysis 1: Comparison: 25% Nitrous Oxide vs Placebo Gas; HAMD-21 at 2 Hours, placebo vs 25% nitrous oxide; Test type: Superiority; p = 0.55, t-test, 2 sided; Mean Difference (Net) = -0.75
Statistical Analysis 2: Comparison: 25% Nitrous Oxide vs Placebo Gas; Change in HAMD-21, 25% nitrous oxide vs placebo at 24 hours; Test type: Superiority; p = 0.47, t-test, 2 sided; Mean Difference (Net) = -1.4
Statistical Analysis 3: Comparison: 50% Nitrous Oxide vs Placebo Gas; HAMD-21 at 2 Hours, placebo vs 50% nitrous oxide; Test type: Superiority; p = 0.49, t-test, 2 sided; Median Difference (Net) = -0.87
Statistical Analysis 4: Comparison: 50% Nitrous Oxide vs Placebo Gas; Change in HAMD-21 at 24 hours, placebo vs 50% nitrous oxide; Test type: Superiority; p = 0.34, t-test, 2 sided; Mean Difference (Net) = -1.9
Statistical Analysis 5: Comparison: 25% Nitrous Oxide vs 50% Nitrous Oxide; Change in HAMD-21 at 2 hours, 25% nitrous oxide vs 50% nitrous oxide; Test type: Superiority; p = 0.94, t-test, 2 sided; Mean Difference (Final Values) = -0.11
Statistical Analysis 6: Comparison: 25% Nitrous Oxide vs 50% Nitrous Oxide; Change in HAMD-21 at 24 hours, 25% nitrous oxide vs 50% nitrous oxide; Test type: Superiority; p = 0.80, t-test, 2 sided; Mean Difference (Net) = -0.5

ADVERSE EVENTS:
Time Frame: 18 weeks
Groups:
- Placebo: Placebo gas: 50% nitrogen(inert), 50% oxygen
- 25% Nitrous Oxide: 25% nitrous oxide, 25% nitrogen, 25% oxygen
- 50% Nitrous Oxide: 50% nitrous oxide, 50% oxygen
Arm/Group | Placebo | 25% Nitrous Oxide | 50% Nitrous Oxide
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 5/22 | 8/20 | 14/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | 25% Nitrous Oxide (N=20) | 50% Nitrous Oxide (N=23)
Haziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Laughing (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Feeling disconnected (Psychiatric disorders) | 1 (1) | 0 (0) | 6 (6)
Feeling high (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Memory gaps (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 4 (4)
Sleepiness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Weakness/heave (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dry Mouth (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Tingling (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Intestinal gas (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Common cold/strep throat (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Stomach virus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Car crash (minor) (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fainting spell (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT03283670/Prot_SAP_000.pdf